CLINICAL TRIAL: NCT06115122
Title: PEPPI Study: Identification of Women at Risk for Placental Dysfunction During the First and Third Trimesters of Pregnancy
Brief Title: PEPPI Study: Identification of Women at Risk for Placental Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Oulu University Hospital (Other)
Collaborators: PerkinElmer, Inc. (Industry); Roche Diagnostics GmbH (Industry); Academy of Finland (Other); Sigrid Jusélius Foundation (Other); Finnish Medical Foundation (Network); University of Oulu (Other)
Responsible Party: Principal Investigator, Jaana Nevalainen, Associate professor, Oulu University Hospital
Other Study IDs: OuluUH_PEPPI
Record Dates: First submitted 2022-11-28; First posted 2023-11-02 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pre-Eclampsia; Intrauterine Growth Restriction; Polycystic Ovary Syndrome; Iron-deficiency; Cardiovascular Diseases; Hypertensive Disorder of Pregnancy; Proteinuria in Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Polycystic Ovary Syndrome; Anemia, Iron-Deficiency; Cardiovascular Diseases; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Blood samples will be taken at first and third trimesters from pregnant women. At birth, blood samples will be taken from umbilical cord, placental samples and umbilical cord samples will be taken also. DNA samples from mothers, fathers and children will be taken. Approximately 900 children will have blood samples at the age of 3 and 6-12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Pre-eclampsia risk group: Approximately 300 women will be enrolled into a risk group according to a pre-eclampsia risk calculator.
  Interventions: Other: Pre-eclampsia screening program
- PCOS group: Women enrolled into study who fulfill ≥2 Rotterdam criteria. Women with PCOS may be included in risk- or control groups.
  Interventions: Other: Pre-eclampsia screening program
- Control group: Approximately 300 women in low risk for pre-eclampsia according to a pre-eclampsia risk calculator.
  Interventions: Other: Pre-eclampsia screening program
- Follow up group: Approximately 2100 women who are not enrolled into risk-, control- or PCOS groups.
  Interventions: Other: Pre-eclampsia screening program
- Children: Mothers and fathers will be asked for permission to follow the child's health information from national registers until the age of 15 years. Approximately 300 children will be recruited to PEPPI-offspring follow up study (including also PCOS offspring).
- Fathers: The role of fathers in the development of pregnancy complications and on the health of the offspring.

INTERVENTIONS:
Other: Pre-eclampsia screening program — Pregnant women will be devided into risk-, control- and PCOS groups according to first trimester screening program.
  Groups: Control group; Follow up group; PCOS group; Pre-eclampsia risk group

SUMMARY:
The main purpose of this study is to evaluate Fetal Medicine Foundation's pre-eclampsia risk calculator using maternal characteristics, first trimester serum placental growth factor (PlGF) and mean arterial pressure (MAP) in a Finnish general population.

Condition or disease: pre-eclampsia, intrauterine growth restriction, polycystic ovary syndrome

DETAILED DESCRIPTION:
According to power calculations, altogether 3000 pregnant women will be recruited into PEPPI-study in Oulu area. Women will be recruited during their first visit to maternity care. Women will have blood samples for study purposes at first and third trimester of pregnancy. Participants will be divided into risk-, control- and polycystic ovary syndrome (PCOS) groups according to pre-eclampsia risk calculation program and questionnaire (PCOS: Rotterdam criteria) (N=300/group). Half of the women in risk- and control groups and all women in PCOS group will have a pregnancy ultrasound scan at 30-32 weeks of gestation. Fathers and children will be recruited at the Oulu University Hospital when the child is born.

Studies within PEPPI-study:

PEPPI-offspring: Children born for those 600 women in risk-, control and PCOS groups who have an extra ultrasound at gestational weeks 30-32 during PEPPI-study and children whose mother developed pre-eclampsia during the pregnancy regardless of her study group during PEPPI-study are recruited into PEPPI-offspring study. PEPPI-offspring study investigates the short- and long-term consequences of placental insufficiency/pre-eclampsia on the health of the children.

PEPPI-PCOS: Investigates pregnancy characteristics of women with PCOS. Women with PCOS form PCOS study group, have additional ultrasound scan at gestational weeks 30-32 and their children are recruited into PEPPI-offspring study.

FERPPI: FERPPI study investigates the possible connection between placental insufficiency and iron deficiency with or without anemia in both pregnant women and their children after birth.

ELIGIBILITY:
Mothers

Inclusion Criteria for PEPPI-study

* Pregnant (first trimester)
* Understands Finnish
* ≥18 years
* Signed informed consent

Exclusion Criteria

* Multiple pregnancy
* Miscarriage/termination of the index pregnancy
* No first trimester blood sampling

Inclusion Criteria for FERPPI-study

* Participates in PEPPI-study (criteria above)
* Blood samples at first and third trimester of pregnancy
* Permits blood sampling from the umbilical cord when the baby is born

Exclusion Criteria

* No first or third trimester blood sampling
* No umbilical cord blood sample after baby is born

Fathers

Inclusion Criteria

* Biological father to the child born for the mother who participated in PEPPI study
* ≥18 years
* Signed informed consent

Exclusion Criteria

• Does not understand Finnish

Children

Inclusion Criteria for PEPPI-study

* Born to mother who participated in PEPPI study
* Signed informed consent from parent(s)

Exclusion Criteria

• No consent from parent(s)

Inclusion Criteria for PEPPI-offspring study • Mother in risk-, control-, or PCOS group during PEPPI-study with ultrasound information at gestational weeks 30-32 or a mother who developed pre-eclampsia during the pregnancy regardless of their study group during PEPPI-study

Exclusion Criteria

• Mother/father declines participation

Inclusion Criteria for FERPPI-study

* Signed informed consent from parent(s)
* Mother has blood samples taken at first and third trimester (iron status)
* Child has blood samples taken at birth and at 3 months of age

Exclusion Criteria

* No consent from parent(s)
* No blood samples from mother
* No blood samples from child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants recruited for PEPPI are pregnant women (females), their partners (males) and babies (female/male).
Study Population: All pregnant women eligible for the study will be invited to participate the study during their first visit to maternity care. Children born to these women and children's fathers will be asked to participate in the study at the labor hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Pregnancy-associated Hypertension and Serious Adverse Outcomes in the Mother or Fetus or Neonate | 20 weeks through discharge following delivery
  Severe hypertension (blood pressure [BP]≥ 160/110) or mild hypertension (BP≥140/90) ≥ 20 weeks gestation in conjunction with one of the following: elevated liver enzymes, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, an indicated preterm birth before 32 weeks of gestation owing to hypertension-related disorders, a fetus that was small for gestational age (SGA, below 3rd percentile) adjusted for sex and race or ethnic group, fetal death after 20 weeks of gestation, or neonatal death
Severe Hypertension | 20 weeks through discharge following delivery
  Women who had severe hypertension only and those who had severe hypertension with elevated liver enzyme levels, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, medically indicated preterm birth, fetal-growth restriction, or fetal death after 20 weeks of gestation, or neonatal death.
Severe or Mild Pregnancy-associated Hypertension With Elevated Liver Enzyme Levels | 20 weeks through discharge following delivery
  Elevated liver enzyme levels are specified as an aspartate aminotransferase level of ≥ 100 U/l. Women who met more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With Thrombocytopenia | 20 weeks through discharge following delivery
  Thrombocytopenia defined as a platelet count of <100 × 109/l. Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With an Elevated Serum Creatinine Level | 20 weeks through discharge following delivery
  Elevated serum creatinine defined as ≥90 µmol/l. Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With an Eclamptic Seizure | 20 weeks through discharge following delivery
  Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With an Indicated Preterm Birth Before 32-34-37 Weeks of Gestation Owing to Hypertension-related Disorders | 20 weeks through discharge following delivery
  Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With a Fetus That Was Small for Gestational Age (Below the - 2 SD) Adjusted for Sex and Race or Ethnic Group | 20 weeks through discharge following delivery
  Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Severe or Mild Pregnancy-associated Hypertension With a Fetal Death After 20 Weeks of Gestation or Neonatal Death | 20 weeks through discharge or prior to discharge following delivery admission
  Women who meet more than one component of the primary outcome are counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Prevalence of high pre-eclampsia risk score in women with PCOS compared to non-PCOS women | at 13 gestational weeks
  Pre-eclampsia risk score is calculated with LifeCycle risk calculation program and a risk of 1:100 or higher is considered as high risk for pre-eclampsia.
11. All the above mentioned outcomes (1-10) in PCOS group compared to non-PCOS group. | 13 gestational weeks through discharge following delivery
  As described above.
The height of the child during the first year of life. | At 0, 3 and 6-12 months of age
  Measurement of height (cm)
The weight of the child during the first year of life. | At 0, 3 and 6-12 months of age
  Measurement of weight (g, kg)
The body mass index (BMI) of the child during the first year of life. | At 0, 3 and 6-12 months of age
  Measurements of height (cm) and weight (kg) combined as BMI (kg/m2)
Basic blood count | At 0, 3 and 6-12 months of age
  B-Hb, B-Leuk, B-Hkr, B-Eryt, E-MCV, E-RDW, E-MCH, E-MCHC, B-Trom
Ferritin | At 0, 3 and 6-12 months of age
Hepcidin | At 0, 3 and 6-12 months of age
Saturation of transferrin | At 0, 3 and 6-12 months of age
Hypersensitive-C-reactive protein | At 0, 3 and 6-12 months of age
Anti-mullerian hormone | At 3 and 6-12 months of age
Cortisol | At 3 and 6-12 months of age
Corticotropin | At 3 and 6-12 months of age
Dehydroepiandrosterone | At 3 and 6-12 months of age
Progesterone | At 3 and 6-12 months of age
Inhibin-B | At 3 and 6-12 months of age
Luteinizing hormone | At 3 and 6-12 months of age
Follicle stimulating hormone | At 3 and 6-12 months of age
Testosterone (boys) | At 3 and 6-12 months of age
Estradioli (girls) | At 3 and 6-12 months of age
Vitamin D | At 3 and 6-12 months of age
Calcium | At 3 and 6-12 months of age
Phosphate | At 3 and 6-12 months of age
Alkaline phosphatase | At 3 and 6-12 months of age
Parathyroid hormone | At 3 and 6-12 months of age
Clinical examination of genitals | At 0, 3 and 6-12 months of age
  Measurement of perineum with centimeters (cm)
Clinical examination of mammary glands | At 3 and 6-12 months of age
  Measurement with millimeters (mm)
Sebum measurement | At 3 and 6-12 months of age
  Measurement is done with Sebumeter ®. The cassette is placed on the skin for a defined length of time and then returned to the aperture. The change in the amount of light transmission represents the sebum content of the tape, which is displayed in units from 0-350.
Heart auscultation with stethoscope. | At 3 and 6-12 months of age
Ultrasound scan of the heart (echo) | At 3 and 6-12 months of age
Birth Weight | At birth
  Grams
Small for Gestational Age | At birth
  A baby whose birth weight is less than the - 2 standard deviations is considered to be small for gestational age (adjusted for sex and race or ethnic group)
Large for gestational age | At birth
  A baby whose birth weight is more than the + 2 standard deviations is considered to be small for gestational age (adjusted for sex and race or ethnic group)
Admission to NICU | Delivery through discharge up to 18 weeks
  NICU denotes neonatal intensive care unit.
Apgar Score ≤3 at 5 Minutes | At birth
Fetal iron deficiency | At birth
  Fetal iron deficiency defined by reticulocyte hemoglobin < 29 pg from umbilical cord blood collected at birth
Iron deficiency during third trimester of pregnancy | At 30-32 weeks of gestation
  Iron deficiency defined as serum ferritin < 30 µg/l at gestational weeks 30-32 with or without anemia defined as Hb ≤ 110 g/l.
Severe iron deficiency during third trimester of pregnancy | At 30-32 weeks of gestation
  Iron deficiency defined as serum ferritin < 15 µg/l at gestational weeks 30-32 with or without anemia defined as Hb ≤ 110 g/l.

SECONDARY OUTCOMES:
Pre-eclampsia (Mild, Severe, HELLP Syndrome, Eclampsia). | 20 weeks through discharge following delivery.
  HELLP denotes hemolytic anemia, elevated liver enzymes, and low platelet count.
Superimposed Pre-eclampsia (Mild, Severe, HELLP Syndrome, Eclampsia). | 20 weeks through discharge following delivery.
  Women with Hypertension before pregnancy week 20. HELLP denotes hemolytic anemia, elevated liver enzymes, and low platelet count.
Pregnancy Associated Hypertension. | 20 weeks through discharge following delivery.
  Women with Hypertension after pregnancy week 20.
Medically Indicated Delivery Because of Hypertension. | 20 weeks through discharge following delivery.
Fetal Weight Estimation under 3rd percentile at gestational weeks 30-32 ultrasound scan. | 30-32 weeks.
Abnormal uterine artery pulsatility index at gestational weeks 30-32 ultrasound scan | At 30-32 weeks.
  According to calculator provided by Fetal Medicine Foundation (https://fetalmedicine.org/research/utpi).
Aspartate Aminotransferase ≥100 U/Liter. | 20 weeks through discharge.
Creatinine ≥90 µmol/l. | 20 weeks through discharge.
Massive postpartum hemorrhage. | From delivery to 24 hours after child birth
  Massive postpartum hemorrhage defined≥ 1000ml blood loss within 24 hours after child birth.
Premature Rupture of Membranes. | From 22nd gestational week until delivery
  If the water breaks before the 37th week of pregnancy, it is called preterm premature rupture of membranes (PPROM).
Placental Abruption. | From 22nd gestational week until delivery
  Defined as the placenta separates from the inner wall of the uterus before birth.
Gestational Diabetes. | From gestation until delivery
  Defined as abnormal glucose tolerance test during pregnancy (≥ 5.3 mmol/l (0 h), ≥ 10.0 mmol/l (1 h) and/or ≥ 8.6 mmol/l (2 h). Treatment either with diet or medicine (metformin and/or insulin therapy).
Cesarean Delivery. | At Birth.
Vacuum Extraction Delivery. | At Birth.
Maternal Death. | During pregnancy or within 42 days after delivery
Postpartum Pulmonary Edema. | Within 42 days after delivery
Hematocrit ≤24% With Transfusion. | Within 42 days after delivery
Maternal Hospital Stay. | Within 42 days after delivery
  Duration of the time spend at the hospital after delivery (measured as days and weeks)
Gestational Age at Delivery. | At Delivery.
Perineal Lacerations. | At Birth.
  Defined as first, second, third or fourth degree lacerations during birth.
Number of Visits to Maternity Health Care During Pregnancy. | From gestation until delivery, on average during 9 months
Number of Visits at Tertiary Maternity Care Hospital. | From gestation until delivery, on average during 9 months
Fetal Death. | From 22nd gestational week until delivery
Neonatal Death. | Birth until 4 weeks' of age
Respiratory Distress Syndrome. | Birth until 4 weeks' of age
Intraventricular Hemorrhage, Grade III or IV. | Birth until 4 weeks' of age
Neonatal sepsis. | Birth until 4 weeks' of age
Necrotizing Enterocolitis. | Birth until 4 weeks' of age
Retinopathy of Prematurity. | Birth until 4 weeks' of age
Neonatal Hospital Stay. | Birth until 18 weeks' of age
Umbilical artery pulsatility index | At 30-32 gestational weeks
  Measured with Doppler ultrasound
Mean cerebral artery pulsatility index | At 30-32 gestational weeks
  Measured with Doppler ultrasound
Ductus venousus pulsatility index | At 30-32 gestational weeks
  Measured with Doppler ultrasound
Fetal weight estimation | At 30-32 gestational weeks
  Measured with ultrasound using fetal BPD, HC, AC and FL measurements (Hadlock)
Amniotic fluid measurement | At 30-32 gestational weeks
  Ultrasound measurements of maximum velocity pocket (cm) and amniotic fluid index (cm)
Estimation of fetal movement during ultrasound scan | At 30-32 gestational weeks
  Estimated as a whole with inspection of body movements, limb movements and breathing movement
Apgar Score ≤7 at 5 minutes. | At birth.
Blood transfusion. | From 22nd pregnancy week until four weeks after delivery
  Defined as red blood cell transfusion received by patient (mother or child).

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Nevalainen, Assoc prof, Principal Investigator — The Wellbeing Services County of North Ostrobothnia
Locations (1):
- The Wellbeing Services County of North Ostrobothnia, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes
Data will deposited into Oulu University Hospital's and Oulu University's data bank.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data is available on request 10 years from study completion
Access Criteria: Data available according to policies of the Oulu University Hospital and Oulu University.

REFERENCES:
- [Background] Maeda K, Naganuma M, Fukuda M, Matsunaga J, Tomita Y. Effect of pituitary and ovarian hormones on human melanocytes in vitro. Pigment Cell Res. 1996 Aug;9(4):204-12. doi: 10.1111/j.1600-0749.1996.tb00110.x. PMID 8948502
- [Background] Bahri Khomami M, Joham AE, Boyle JA, Piltonen T, Silagy M, Arora C, Misso ML, Teede HJ, Moran LJ. Increased maternal pregnancy complications in polycystic ovary syndrome appear to be independent of obesity-A systematic review, meta-analysis, and meta-regression. Obes Rev. 2019 May;20(5):659-674. doi: 10.1111/obr.12829. Epub 2019 Jan 23. PMID 30674081
- [Background] Becker M, Hesse V. Minipuberty: Why Does it Happen? Horm Res Paediatr. 2020;93(2):76-84. doi: 10.1159/000508329. Epub 2020 Jun 29. PMID 32599600
- [Background] Binder NK, Evans J, Salamonsen LA, Gardner DK, Kaitu'u-Lino TJ, Hannan NJ. Placental Growth Factor Is Secreted by the Human Endometrium and Has Potential Important Functions during Embryo Development and Implantation. PLoS One. 2016 Oct 6;11(10):e0163096. doi: 10.1371/journal.pone.0163096. eCollection 2016. PMID 27711226
- [Background] Chockalingam UM, Murphy E, Ophoven JC, Weisdorf SA, Georgieff MK. Cord transferrin and ferritin values in newborn infants at risk for prenatal uteroplacental insufficiency and chronic hypoxia. J Pediatr. 1987 Aug;111(2):283-6. doi: 10.1016/s0022-3476(87)80088-4. PMID 3612404
- [Background] Dewey KG, Oaks BM. U-shaped curve for risk associated with maternal hemoglobin, iron status, or iron supplementation. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1694S-1702S. doi: 10.3945/ajcn.117.156075. Epub 2017 Oct 25. PMID 29070565
- [Background] Duley L. The global impact of pre-eclampsia and eclampsia. Semin Perinatol. 2009 Jun;33(3):130-7. doi: 10.1053/j.semperi.2009.02.010. PMID 19464502
- [Background] Duley L, Henderson-Smart DJ, Meher S, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004659. doi: 10.1002/14651858.CD004659.pub2. PMID 17443552
- [Background] Guy GP, Leslie K, Diaz Gomez D, Forenc K, Buck E, Khalil A, Thilaganathan B. Implementation of routine first trimester combined screening for pre-eclampsia: a clinical effectiveness study. BJOG. 2021 Jan;128(2):149-156. doi: 10.1111/1471-0528.16361. Epub 2020 Jul 1. PMID 32613730
- [Background] Henley D, Brown S, Pennell C, Lye S, Torpy DJ. Evidence for central hypercortisolism and elevated blood pressure in adolescent offspring of mothers with pre-eclampsia. Clin Endocrinol (Oxf). 2016 Oct;85(4):583-9. doi: 10.1111/cen.13092. Epub 2016 May 26. PMID 27144974
- [Background] Kalousova M, Muravska A, Zima T. Pregnancy-associated plasma protein A (PAPP-A) and preeclampsia. Adv Clin Chem. 2014;63:169-209. doi: 10.1016/b978-0-12-800094-6.00005-4. PMID 24783354
- [Background] Koster MP, de Wilde MA, Veltman-Verhulst SM, Houben ML, Nikkels PG, van Rijn BB, Fauser BC. Placental characteristics in women with polycystic ovary syndrome. Hum Reprod. 2015 Dec;30(12):2829-37. doi: 10.1093/humrep/dev265. Epub 2015 Oct 25. PMID 26498178
- [Background] Nevalainen J, Korpimaki T, Kouru H, Sairanen M, Ryynanen M. Performance of first trimester biochemical markers and mean arterial pressure in prediction of early-onset pre-eclampsia. Metabolism. 2017 Oct;75:6-15. doi: 10.1016/j.metabol.2017.07.004. Epub 2017 Jul 18. PMID 28964327
- [Background] Nevalainen J, Skarp S, Savolainen ER, Ryynanen M, Jarvenpaa J. Intrauterine growth restriction and placental gene expression in severe preeclampsia, comparing early-onset and late-onset forms. J Perinat Med. 2017 Oct 26;45(7):869-877. doi: 10.1515/jpm-2016-0406. PMID 28593875
- [Background] O'Gorman N, Wright D, Rolnik DL, Nicolaides KH, Poon LC. Study protocol for the randomised controlled trial: combined multimarker screening and randomised patient treatment with ASpirin for evidence-based PREeclampsia prevention (ASPRE). BMJ Open. 2016 Jun 28;6(6):e011801. doi: 10.1136/bmjopen-2016-011801. PMID 27354081
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Santos DCC, Angulo-Barroso RM, Li M, Bian Y, Sturza J, Richards B, Lozoff B. Timing, duration, and severity of iron deficiency in early development and motor outcomes at 9 months. Eur J Clin Nutr. 2018 Mar;72(3):332-341. doi: 10.1038/s41430-017-0015-8. Epub 2017 Nov 6. PMID 29235557
- [Background] Shanmugalingam R, Hennessy A, Makris A. Aspirin in the prevention of preeclampsia: the conundrum of how, who and when. J Hum Hypertens. 2019 Jan;33(1):1-9. doi: 10.1038/s41371-018-0113-7. Epub 2018 Sep 19. PMID 30232399
- [Background] Shao J, Lou J, Rao R, Georgieff MK, Kaciroti N, Felt BT, Zhao ZY, Lozoff B. Maternal serum ferritin concentration is positively associated with newborn iron stores in women with low ferritin status in late pregnancy. J Nutr. 2012 Nov;142(11):2004-9. doi: 10.3945/jn.112.162362. Epub 2012 Sep 26. PMID 23014493
- [Background] Tal R, Seifer DB, Grazi RV, Malter HE. Follicular fluid placental growth factor is increased in polycystic ovarian syndrome: correlation with ovarian stimulation. Reprod Biol Endocrinol. 2014 Aug 20;12:82. doi: 10.1186/1477-7827-12-82. PMID 25141961
- [Background] Tan MY, Wright D, Syngelaki A, Akolekar R, Cicero S, Janga D, Singh M, Greco E, Wright A, Maclagan K, Poon LC, Nicolaides KH. Comparison of diagnostic accuracy of early screening for pre-eclampsia by NICE guidelines and a method combining maternal factors and biomarkers: results of SPREE. Ultrasound Obstet Gynecol. 2018 Jun;51(6):743-750. doi: 10.1002/uog.19039. Epub 2018 Mar 14. PMID 29536574
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Yliniemi A, Nurkkala MM, Kopman S, Korpimaki T, Kouru H, Ryynanen M, Marttala J. First trimester placental retinol-binding protein 4 (RBP4) and pregnancy-associated placental protein A (PAPP-A) in the prediction of early-onset severe pre-eclampsia. Metabolism. 2015 Apr;64(4):521-6. doi: 10.1016/j.metabol.2014.12.008. Epub 2014 Dec 26. PMID 25633269
- See also: PEPPI-study's webpage — http://www.peppitutkimus.fi